CLINICAL TRIAL: NCT00591487
Title: Safety and Efficacy of Lidocaine Infiltration in Suction Assisted Lipectomy With Tumescent Technique. A Randomized, Double Blinded, Controlled Trial.
Brief Title: Safety and Efficacy of Lidocaine Infiltration in Suction Assisted Lipectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital Militar de Santiago (Other)
Responsible Party: Stefan Danilla, MD, MSc, Hospital Militar de Santiago
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HMS-LIPO-001; HMS-LIPO-001
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
Keywords: suction; assisted; lipectomy; liposuction; contour; cosmetic; plastic; surgery; Klein; tumescent; technique; Healthy women wanting Suction Assisted Lipectomy
MeSH Terms: conditions — Helping Behavior | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator): Infiltration with 0.9% saline+1:1,000,000 epinephrine+0.06% Lidocaine
  Interventions: Drug: Lidocaine
- II (Placebo Comparator): Infiltration with 0.9% saline+1:1,000,000 epinephrine
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Subcutaneous infiltration with Active/Placebo solutions with tumescent technique previous to suction assisted lipectomy. Patient abdomen and back will be divided in 4 zones anterior and posterior, one side (left or right) will be infiltrated with active solution and the other with placebo. The allocation of the side will be made with random numbers.

SUMMARY:
RCT of S/E of lidocaine infiltration in tumescent technique.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* I or II of the Classification of the American Society of Anesthesiologists.
* Completed high school.
* Between 18 and 40 years old
* At least suction of entire abdomen and back
* Body mass index between 20 and 27
* Accept written informed consent

Exclusion Criteria:

* Associated surgery
* Hypersensibility to (Cefazolin or Clindamycin, Lidocaine, Ketorolac, Morphine, Remifentanyl, Propofol, Tramadol).
* Pregnancy
* Previous surgery to abdominal wall or back, including cesarean.
* Abdominal wall hernia
* Previous liposuction
* Active psychosis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Pain (VSA) | 1, 6, 12, 18 and 24 post operative hours

SECONDARY OUTCOMES:
Rescue medication | 1, 6, 12, 15 and 24 hours postoperative
Nausea, emesis, arrythmia, seizures, arrest, shock, death. | 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Danilla, MD, MSc, Principal Investigator — Hospital Militar de Santiago; Guillermo Israel, MD, Study Chair — Hospital Militar de Santiago; Montserrat Fontbona, MD, Study Chair — Hospital Militar de Santiago; Rodrigo Cabello, MD, Study Director — Hospital Militar de Santiago
Locations (1):
- Hospital Militar de Santiago, Santiago, RM, Chile

REFERENCES:
- [Background] Kaplan B, Moy RL. Comparison of room temperature and warmed local anesthetic solution for tumescent liposuction. A randomized double-blind study. Dermatol Surg. 1996 Aug;22(8):707-9. doi: 10.1111/j.1524-4725.1996.tb00621.x. PMID 8780763
- [Background] Yang CH, Hsu HC, Shen SC, Juan WH, Hong HS, Chen CH. Warm and neutral tumescent anesthetic solutions are essential factors for a less painful injection. Dermatol Surg. 2006 Sep;32(9):1119-22; discussion 1123. doi: 10.1111/j.1524-4725.2006.32254.x. PMID 16970691
- [Background] Rubin JP, Bierman C, Rosow CE, Arthur GR, Chang Y, Courtiss EH, May JW Jr. The tumescent technique: the effect of high tissue pressure and dilute epinephrine on absorption of lidocaine. Plast Reconstr Surg. 1999 Mar;103(3):990-6; discussion 997-1002. PMID 10077095
- [Background] Rubin JP, Xie Z, Davidson C, Rosow CE, Chang Y, May JW Jr. Rapid absorption of tumescent lidocaine above the clavicles: a prospective clinical study. Plast Reconstr Surg. 2005 May;115(6):1744-51. doi: 10.1097/01.prs.0000161678.10555.53. PMID 15861085
- [Derived] Danilla S, Fontbona M, de Valdes VD, Dagnino B, Sorolla JP, Israel G, Searle S, Norambuena H, Cabello R. Analgesic efficacy of lidocaine for suction-assisted lipectomy with tumescent technique under general anesthesia: a randomized, double-masked, controlled trial. Plast Reconstr Surg. 2013 Aug;132(2):327-332. doi: 10.1097/PRS.0b013e3182958b20. PMID 23897332
- See also: Related Info — http://www.hosmil.cl